CLINICAL TRIAL: NCT03372291
Title: Randomized Study of a Psychological Intervention Mobile Application (App) to Promote Coping in Patients With Acute Myeloid Leukemia (AML)
Brief Title: Psychological Intervention Mobile App for Patients With AML
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-542
Record Dates: First submitted 2017-12-09; First posted 2017-12-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological app (Experimental): Psychological intervention consist of four components
  * Supportive psychotherapy interventions to help patients deal with the initial shock of diagnosis, cope with the loss of independence and abrupt life disruptions, and provide validation and reassurance;
  * Psychoeducation to manage expectations and enhance preparedness for extended hospitalization and mobilize social supports;
  * Psychosocial skill-building to promote effective coping strategies and facilitate acceptance while living with uncertainty;
  * Self-care to promote positive health behaviors and enhance patients' sense of control especially as they transition from the hospital to outpatient care.
  * The psychological intervention will consist of four sessions (20-25 minutes each) that patients will start during their first week of admission for intensive chemotherapy and continue weekly
  Interventions: Other: Psychological intervention
- Usual Care (Active Comparator): * Participants receiving usual care will not have access to the psychological intervention app. -They will receive usual leukemia care with all the supportive care measures instituted by the leukemia team.
  * Patients in usual care will also meet with the leukemia social worker based on their request or at the discretion of the treating leukemia team
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Usual Care — Usual leukemia care with all the supportive care measures instituted by the leukemia team
  Arms: Usual Care
Other: Psychological intervention — Psychological intervention is focused on educating patients about leukemia and how to cope with its treatment
  Arms: Psychological app

SUMMARY:
This research study is evaluating the impact of a psychological intervention mobile application (app) on the quality of life, mood, and symptoms of patients with acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
Patients with a new diagnosis of AML often confront a sudden and life-threatening diagnosis, requiring an immediate disruption of their life and an urgent 4-6 week hospitalization to initiate intensive chemotherapy. During this hospitalization, they endure substantial physical symptoms due to the side-effects of intensive chemotherapy, which negatively impacts their quality of life (QOL). Patients with AML also experience significant psychological distress as they struggle with the abrupt onset of illness, uncertainty regarding their prognosis, physical and social isolation during their hospitalization, and complete loss of independence. The study doctors want to know if the use of a mobile application (app) focused on helping patients cope with the diagnosis and treatment can reduce the distressing symptoms and improve the their quality of life and care.

The main purpose of this research study is see if a mobile app is feasible to use for patients with new diagnosis of AML and is acceptable to them. The study will also compare two types of care - standard leukemia care and standard leukemia care with the mobile app to see which is better for improving the experience of patients newly diagnosed with AML undergoing treatment.

The purpose of this research study is to find out whether using the mobile app that is focused on educating patients about leukemia and how to cope with its treatment can improve the physical and psychological symptoms that patients experience during hospitalization for their leukemia care. Using this research, the study doctors hope to find out the best way to help patients cope with their diagnosis and treatment for acute myeloid leukemia.

The study will use questionnaires to measure patient's quality of life, physical symptoms, mood, and the participant sense of control over their situation. Study questionnaires will be completed in the hospital or clinic with assistance provided as needed. The participants will also have the option of completing these questionnaires remotely through a secure web link or through a mailed paper copy

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years).
* New diagnosis of acute myeloid leukemia.
* Admitted to Massachusetts General Hospital for intensive induction chemotherapy requiring 4-6-week hospitalization.
* The ability to provide informed consent.
* Ability to comprehend and speak English.

Exclusion Criteria:

* Significant uncontrolled psychiatric disorder (psychotic disorder, bipolar disorder,
* Major depression) or other co-morbid disease (dementia, cognitive impairment), which the treating clinician believes prohibits the ability to participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Feasibility based on proportion of subjects enrolled and completing the app modules | 2 years
  The intervention will be deemed feasible if at least 60% of eligible patients are enrolled in the study and for those enrolled, they must complete at least 60% of the intervention modules.

SECONDARY OUTCOMES:
Mood as measured by the Hospital Anxiety and Depression Scale (HADS) | up to day +40 after intensive chemotherapy
  Compare patient mood as measured by the Hospital Anxiety and Depression Scale (HADS) between the mobile app intervention and standard leukemia care. The HADS includes a depression and anxiety subscales (range 0 to 21) with higher scores indicating higher level of distress
Patient depression syndrome as measured by the Patient-Health Questionnaire-9 (PHQ-9) | up to day +40 after intensive chemotherapy
  Compare patient depression symptoms as measured by the Patient Health Questionnaire (PHQ-9) between the mobile app intervention and standard leukemia care. The PHQ-9 has a score range of 0 to 27, with higher scores indicating worse depression symptoms.
Quality of life as measured by the Functional Assessment of Cancer Therapy- Leukemia (FACT-Leuk) | up to day +40 after intensive chemotherapy
  Compare patient QOL as measured by the Functional Assessment of Cancer Therapy (FACT-Leukemia) between the mobile app intervention and standard leukemia care. The FACT-Leukemia score ranges from 0 to 176 with higher scores indicating better quality of life.
Symptom burden as measured by the Edmonton Symptom Assessment Scale (ESAS) | up to day +40 after intensive chemotherapy
  Compare patient symptom burden as measured by the Edmonton Symptom Assessment Scale (ESAS) between the mobile app intervention and standard leukemia care. ESAS scores range from 0 to 100 with higher scores indicating worse symptom burden.
Patient self-efficacy as measured by the Cancer Self-Efficacy Scale (CASE) | up to day +40 after intensive chemotherapy
  Compare patient self-efficacy as measured by CASE between the mobile app intervention and standard leukemia care. The CASE has a score range of 0 to 170 with higher scores indicating a better sense of self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jensen-Battaglia M, Sohn MB, Consagra W, Wang Y, Zhang Z, LoCastro M, Davis J, Buettner K, Mortaz S, El-Jawahri AR, Loh KP. Trajectories of physical well-being among adults with acute myeloid leukemia. Blood Adv. 2024 Jun 11;8(11):2612-2621. doi: 10.1182/bloodadvances.2023011804. PMID 38429079
- [Derived] El-Jawahri A, Luskin MR, Greer JA, Traeger L, Lavoie M, Vaughn DM, Andrews S, Yang D, Boateng KY, Newcomb RA, Ufere NN, Fathi AT, Hobbs G, Brunner A, Abel GA, Stone RM, DeAngelo DJ, Wadleigh M, Temel JS. Psychological mobile app for patients with acute myeloid leukemia: A pilot randomized clinical trial. Cancer. 2023 Apr 1;129(7):1075-1084. doi: 10.1002/cncr.34645. Epub 2023 Jan 18. PMID 36655338